CLINICAL TRIAL: NCT07366372
Title: The Efficacy of Taurolidine Containing Lock Solution for Prevention of Central Venous Catheter Infection in ICU Patients
Brief Title: Efficacy of Taurolidine Containing Lock Solution for Prevention of Central Venous Catheter Infection in ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Doaa Kelany Zakaria Ibrahim, Assistant Lecturer of Anesthesiology, Intensive Care and Pain Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264MD73/4/23
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Taurolidine; Lock Solution; Prevention; Central Venous Catheter Infection; Intensive Care Unit
MeSH Terms: interventions — Sodium Chloride; Tigecycline; Heparin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Placebo Comparator): Central venous catheters (CVCs) were locked with 2ml saline as a control group.
  Interventions: Drug: Saline
- Group II (Experimental): Central venous catheters (CVCs) were locked with 2ml of a solution comprising tigecycline 5mg/ml and heparin 500 IU/ml.
  Interventions: Drug: Tigecycline and heparin
- Group III (Experimental): Central venous catheters (CVCs) were locked with 2ml of a solution containing taurolidine-citrate-heparin (1.35% taurolidine, 4% citrate, and 500 IU/ml heparin).
  Interventions: Drug: Taurolidine-citrate-heparin

INTERVENTIONS:
Drug: Saline — Central venous catheters (CVCs) were locked with 2ml saline as a control group.
  Arms: Group I
Drug: Tigecycline and heparin — Central venous catheters (CVCs) were locked with 2ml of a solution comprising tigecycline 5mg/ml and heparin 500 IU/ml.
  Arms: Group II
Drug: Taurolidine-citrate-heparin — Central venous catheters (CVCs) were locked with 2ml of a solution containing taurolidine-citrate-heparin (1.35% taurolidine, 4% citrate, and 500 IU/ml heparin).
  Arms: Group III

SUMMARY:
This study aimed to assess effectiveness of a taurolidine based lock solution in preventing the infections of central venous catheter (CVC) in intensive care unit (ICU) cases.

DETAILED DESCRIPTION:
The central venous catheter (CVC) is highly frequent in the intensive care unit (ICU), with an average use rate between 32% and 80% among adult ICU patients. The utilization of CVC in ICUs has escalated over the past decade, accompanied by a corresponding increase in problems related to their usage.

Taurolidine is a nontoxic substance having antibacterial impacts counter to mutually gram-positive and -negative bacteria, additionally to fungus. It decreases biofilm development and doesn't develop resistance to antibiotics, since it serves as an antiseptic rather than an antibiotic Consequently, it may function as a locking mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years.
* Both genders.
* Patients admitted to the intensive care unit (ICU) requiring central venous catheter insertion.

Exclusion Criteria:

* Cases with active infections, hemorrhage or bleeding disorders, infections within insertion place.
* History of allergy to taurolidine, tigecycline, heparin, and citrate.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Positive bacterial growth | 30 days after the procedure
  Positive bacterial growth of a swab was recorded.

SECONDARY OUTCOMES:
Assessment of catheter-related bloodstream infection | 30 days after the procedure
  Assessment of catheter-related bloodstream infection was recorded.
Assessment of central venous catheter infection | 30 days after the procedure
  Assessment of central venous catheter (CVC) infection was recorded.
Lenght of intensive care unit stay | 30 days after the procedure
  Lenght of intensive care unit (ICU) stay was recorded.
Incidence of mortality | 30 days after the procedure
  Incidence of mortality was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.